CLINICAL TRIAL: NCT07054580
Title: Knowledge and Awareness of Instruments Sterilization Protocols Among Healthcare Workers in Operation Theater
Status: Active, not recruiting | Type: Observational
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Other Study IDs: MSAHSW/Batch-Fall23/923
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Awareness, Anesthesia
MeSH Terms: conditions — Intraoperative Awareness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: knowledge and awareness — Focus on the level of knowledge and awareness regarding instrument sterilization protocols among healthcare workers in the operation theater.

SUMMARY:
In the medical field, the sterilization of instruments is a crucial component of any surgical procedure. It's important for healthcare workers to have a fundamental understanding of how to properly sterilize and disinfect instruments and medical devices. Despite its importance, there are often gaps in the knowledge and adherence to sterilization protocols among healthcare workers, which can lead to increased risks of healthcare-associated infections.

DETAILED DESCRIPTION:
This research aims to assess healthcare workers' awareness and understanding of sterilization practices, identify challenges they face, and propose strategies for improving sterilization practices in healthcare environments.

ELIGIBILITY:
Inclusion Criteria:

* All OT Staff is included
* Both Male and Female Gender
* Age 20 or Above

Exclusion Criteria:

* other than OT staff

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A questionnaire will be developed to assess the knowledge and awareness levels of various healthcare workers. Participants will be answered all questions and submitted their responses via an online link. The study will be conducted over 4 months and included 30 questions, with 15 focused on knowledge and 15 on awareness
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Knowledge and Awareness Scale self | 12 Months
  A questionnaire will be developed to assess the knowledge and awareness levels of various healthcare workers. Participants will be answered all questions and submitted their responses via an online link. The study will be conducted over 4 months and included 30 questions, with 15 focused on knowledge and 15 on awareness

CONTACTS AND LOCATIONS:
Locations (1):
- Shalamar Hospital Mughalpura, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No